CLINICAL TRIAL: NCT05080543
Title: Recruitment of Microcirculation Using Albumin 20% and Terlipressin in Patients With Septic Shock: a Randomized Controlled Double-blinded Study.
Brief Title: Microcirculation Recruitment Using Albumin 20% and Terlipressin in Septic Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amany Mousa Salama Muhammed (Other)
Responsible Party: Sponsor-Investigator, Amany Mousa Salama Muhammed, CairoU, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Microcirculation septic shock
Record Dates: First submitted 2021-09-29; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Septic Shock
Keywords: Microcirculation; Terlipressin; Human Albumin 20%
MeSH Terms: conditions — Shock, Septic | interventions — Albumins; Terlipressin; Microcirculation

STUDY DESIGN:
Intervention Model Description: a randomized controlled and double-blinded
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group AT (Active Comparator): will receive a bolus of albumin (1gm/kg) and terlipressin loading dose of 1 mg over 20 minutes followed by infusion at rate (2 μ g/kg/h)
  Interventions: Drug: Albumin 20% and terlipressin
- Controlled (Placebo Comparator): will receive the routine management of septic shock patients as culture-based IV antibiotics, IV fluids and intropic support plus a placebo (as lactated ringer solution in the same infusion rates for blinding).
  Interventions: Drug: Albumin 20% and terlipressin

INTERVENTIONS:
Drug: Albumin 20% and terlipressin — Evaluation the effect of adding 20% HSA and terlipressin on microvascular ﬂow index (MFI), flow heterogeneity index, total vessel density (TVD), and perfused vessel density (PVD) in comparison to the standard care in patient with septic shock.
  Other Names: Microcirculation

SUMMARY:
The aim of this study is to evaluate the effect of combining HSA 20% and terlipressin on the microcirculation in patients with septic shock using the following;-

* Microcirculation recruitment by Cytocam-IDF.
* Cardiac output by LiDCOrapid.
* Measuring serum lactate level.

DETAILED DESCRIPTION:
Sepsis is one of the major medical problems and is responsible for high morbidity and mortality. Surviving Sepsis Campaign Guideline 2016 introduced 3-hours and 6-hours bundles in management of septic shock. The 2018 update of the Surviving Sepsis Campaign guidelines introduced the 'Hour-1 Bundle' which recommends treatment with intravenous fluids, measurement of serum lactate concentration as a marker of illness severity, administration of vasopressors, obtaining blood cultures and administering broad-spectrum antibiotics, all within the first hour.

The usual targets for resuscitation of patients with septic shock are the macro-circulatory parameters such as mean arterial blood pressure and heart rate; however, it is believed that restoration of microcirculatory parameters is not sufficient to avoid organ failure unless it was associated with improved microcirculatory perfusion. The loss of coherence between macro- and micro-circulatory parameters increases the need to evaluate the microcirculatory blood flow. So impaired microvascular perfusion is increasingly recognized as a major determinant of tissue hypoxia during sepsis and is a key factor in the pathogenesis of sepsis-induced organ failure.

Fluid resuscitation is recommended to be initiated immediately and completed within the first hour. Guidelines recommend at least a 30-mL/kg bolus of crystalloid fluid as the initial resuscitation. Crystalloid is the fluid of choice for initial resuscitation and subsequent intra-vascular volume replacement in patients with sepsis and septic shock.

Albumin in addition to crystalloids is suggested when patients require a substantial amount of crystalloids. Although the guidelines make no recommendation regarding which concentration of albumin should be used, 5% albumin is most commonly used in patients with hypovolemia to administer as much volume as possible.

In 2016, a study showed that in a rat model of normotensive endotoxemia, the infusion of 4% or 20% Human Serum Albumin "HSA" restored microvascular perfusion in otherwise unresuscitated animals. A more stable microvascular improvement noticed with 20% HSA.

Sepsis is also characterized by an enhanced activation of inflammatory and oxidative stress pathways, which leads to endothelial dysfunction and vascular hyporeactivity.

For its ability to counteract oxidative and nitrosative stress, albumin may represent not only a plasma expander but also an endothelium-modulating agent. In an experimental rodent model of endotoxemia, (HSA) prevented endothelial dysfunction and vascular hyporeactivity.

In patients with septic shock requiring vasopressors, a targeted mean arterial pressure "MAP" of 65 mm Hg within the first hour is recommended. Norepinephrine is the recommended first-line vasopressor in septic shock. If MAP is not maintained at 65 mm Hg or greater with norepinephrine alone or if the norepinephrine dose needs to be decreased, either vasopressin (up to 0.03 unit/minute) or epinephrine can be added to norepinephrine. Although norepinephrine is widely regarded as the first-line vasoactive medication in sepsis, literature continues to debate whether the early addition of vasopressin should be common practice.

Terlipressin is a synthetic analogue of vasopressin which has greater selectivity for the V1 receptor that cause vascular smooth muscle vasoconstriction in response to vasopressin and thus could be associated with fewer side effects than vasopressin.

In 2016 a study showed that terlipressin therapy was associated with good improvement in hemodynamic variables and kidney functions more than adrenaline in patients with refractory septic shock despite adequate fluid resuscitation and the use of norepinephrine.

No data was found on effect of combination of albumin and terlipressin on microcirculation in septic patients.

This study aims to investigate the effect of this combination on microcirculation using Cytocam-IDF (incident dark-field illumination), Braedius.

ELIGIBILITY:
Inclusion Criteria:

* The presence of septic shock meeting all of the following criteria less than 24 hours:-

  1. Clinically possible or probable or microbiologically confirmed infection taking into account the definitions of the "International Sepsis Forum (ISF)"
  2. Despite adequate volume therapy, vasopressors are required to maintain mean arterial pressure (MAP) ≥ 65 mm Hg.
  3. Serum lactate level > 2 mmol/l (18 mg/dl) despite adequate volume therapy.

Exclusion Criteria:

* Patients who failed to achieve target MAP despite adequate resuscitation with fluids and maximum dose of noreadrenaline.
* Acute coronary artery disease or underlying cardiac dysfunction [cardiac index (CI) <2.2 l/min/m 2 ].
* Severe liver disease (Child-Pugh grade C)
* Chronic renal failure.
* Known hypersensitivity to Norepinephrine, terlipressin and human albumin.
* Those having Raynaud's phenomenon, or a vasospastic diathesis and
* Other causes of shock e.g.; hemorrhagic hypovolaemia, cardiogenic shock, anaphylactic shock, neurogenic shock.
* Pregnant patients and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Mean Flow Index 6hs | 6 hrs
  Determination the degree the mean flow index (MFI) 6 hrs after administration albumin and terlipressin in patient with septic shock

SECONDARY OUTCOMES:
Mean Flow Index 24hs | 24 hs
  Determination the degree the mean flow index (MFI) 24 hrs after administration albumin and terlipressin in patient with septic shock.